CLINICAL TRIAL: NCT03930264
Title: A Single Centre, Two Period Crossover Study to Assess the Bioequivalence of an Oral Azathioprine Suspension 10 mg/mL (Jayempi™) Versus Oral Azathioprine Tablet 50mg (Imurek®) in at Least 30 Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence of Azathioprine Suspension 10 mg/mL (Jayempi) Versus Azathioprine Tablet 50mg (Imurek®)
Acronym: AZA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Laboratories Limited (Industry)
Collaborators: Medicines Evaluation Unit Ltd (Industry); Syne Qua Non Limited (Industry); Alderley Analytical Ltd. (Industry); Black County Pathology Services (Other); Diamond Pharma Services Regulatory Affairs Consultancy (Other); Boyd Consultants (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: INV691
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Therapeutic Equivalency
MeSH Terms: interventions — Azathioprine; Suspensions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imurek®, (Active Comparator): Generic name : Azathioprine Trade name : Imurek® 50mg tablet Dosage form : Tablet containing 50 mg azathioprine Dose : 1 x Imurek 50mg Tablet per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Aspen Pharma Trading Limited, Dublin, Ireland Country of origin : Ireland
  Interventions: Drug: Azathioprine 50Mg Tab
- Jayempi™ (Experimental): Generic name : Azathioprine
  Trade name : (Jayempi™) 10 mg/ mL Oral solution Dosage form : Oral suspension containing 10 mg/mL Azathioprine Dose : 1 x 5mL (50 mg) of Jayempi™ Oral Suspension 10mg/mL per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Nova Laboratories Ltd. Country of origin : Leicester, UK
  Interventions: Drug: Azathioprine 10mg/mL oral suspension

INTERVENTIONS:
Drug: Azathioprine 50Mg Tab — tablet
  Other Names: Imurek
  Arms: Imurek®,
Drug: Azathioprine 10mg/mL oral suspension — oral suspension
  Other Names: Jayempi
  Arms: Jayempi™

SUMMARY:
A single center, single dose, open-label, randomized, two period crossover study to assess the bioequivalence of an oral azathioprine suspension 10 mg/mL (Jayempi™) versus oral azathioprine tablet 50mg (Imurek®, Aspen Pharma Trading Limited, Dublin, Ireland.) in at least 30 healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
This will be a single-dose, open-label, randomised, two-period crossover study with orally administered 1 x 5mL (50 mg) of Jayempi™ Oral Suspension 10mg/mL versus oral azathioprine tablet 50mg (Imurek®, Aspen Pharma Trading Limited, Dublin, Ireland) on two separate occasions conducted under fasting conditions in healthy male and female subjects at a single study centre.

The study will comprise:

* Thiopurine methyltransferase (TPMT) testing;
* Screening period of maximum 28 days
* Two treatment periods (each of which will include a PK profile period of 12 hours) separated by a wash-out period of at least 3 calendar days (minimum number of days based on half-life of the analyte) and maximum of 14 calendar days between consecutive administrations of the IMP
* A post-study visit 7-10 days after the last dose of the last treatment period of the study.

Subjects will be randomly assigned to treatment sequence, prior to the first administration of IMP.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers.
* No significant medical history or conditions that may interfere with the study.
* Adequate contraception.

Exclusion Criteria:

* Volunteers who may be likely to have the inherited mutated NUDT15.
* Subjects with a deficient, low or intermediate TPMT enzyme activity.
* Disease that may interfere with the safety of the participant or the study outcome measures.
* Participants who want to procreate in the next 6 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naimat Khan, MD, Principal Investigator — Medicines Evaluation Unit
Locations (2):
- United Kingdom (2):
  - Nova Laboratories Limited, Leicester, Leicestershire
  - Medicines Evaluation Unit Ltd Southmoor Road, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cross Over
Groups:
- Imurek®, First: Generic name : Azathioprine Trade name : Imurek® 50mg tablet Dosage form : Tablet containing 50 mg azathioprine Dose : 1 x Imurek 50mg Tablet per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Aspen Pharma Trading Limited, Dublin, Ireland Country of origin : Ireland
  Azathioprine: tablet
- Jayempi™ First: Generic name : Azathioprine
  Trade name : (Jayempi™) 10 mg/ mL Oral solution Dosage form : Oral suspension containing 10 mg/mL Azathioprine Dose : 1 x 5mL (50 mg) of Jayempi™ Oral Suspension 10mg/mL per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Nova Laboratories Ltd. Country of origin : Leicester, UK
  Azathioprine: oral suspension
Period: Overall Study
Arm/Group | Imurek®, First | Jayempi™ First
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Jayempi™, First: Generic name : Azathioprine
  Trade name : (Jayempi™) 10 mg/ mL Oral solution Dosage form : Oral suspension containing 10 mg/mL Azathioprine Dose : 1 x 5mL (50 mg) of Jayempi™ Oral Suspension 10mg/mL per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Nova Laboratories Ltd. Country of origin : Leicester, UK
  Azathioprine: oral suspension
- Total: Total of all reporting groups
Arm/Group | Imurek®, First | Jayempi™, First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 40.8 (9.00) | 33.5 (9.61) | 37 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The maximum (peak) plasma concentration assesses the rate of drug absorption
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Imurek: Tablet formulation
- Jayempi™: Liquid formulation
Arm/Group | Imurek | Jayempi™
Number analyzed (Participants) | 29 | 29
ng/mL | 15.49 (67.1) | 17.35 (54.4)
Statistical Analysis 1: Comparison: Imurek vs Jayempi™; Test type: Equivalence — For bioequivalence, the 90% CIs of the geometric mean ratio of Cmax for tablet and suspension were required to be within the 80 to 125% range; p = 0.3008, ANOVA; Odds Ratio (OR) = 1.12, 90% CI 2-sided [0.93 to 1.35]

2. Primary Outcome: AUC0-t
Description: Area under the curve time=0 hours to t hours
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Imurek | Jayempi™
Number analyzed (Participants) | 29 | 29
h.ng/mL | 17.10 (33.8) | 18.17 (32.1)
Statistical Analysis 1: Comparison: Imurek vs Jayempi™; Test type: Equivalence — For bioequivalence, the 90% CIs of the geometric mean ratio of AUC0-τ for tablet and suspension were required to be within the 80 to 125% range; p = 0.1061, ANOVA; Ratio = 1.06, 90% CI 2-sided [1.00 to 1.13]

3. Primary Outcome: AUC0-∞
Description: Area under to curve from time=0 hours to infinity
Time Frame: 18 hours
Measure: Mean (Standard Deviation); unit: h.ng/mL
Arm/Group | Imurek | Jayempi™
Number analyzed (Participants) | 23 | 26
h.ng/mL | 17.71 (27.1) | 18.96 (31.6)
Statistical Analysis 1: Comparison: Imurek vs Jayempi™; Test type: Equivalence — For bioequivalence, the 90% CIs of the geometric mean ratio of AUC0-∞ for tablet and suspension were required to be within the 80 to 125% range; p = 0.5696, ANOVA; Ratio = 1.02, 90% CI 2-sided [0.96 to 1.09]

ADVERSE EVENTS:
Time Frame: AEs were collected up to the end of the follow-up period (up to 10 days after Treatment period 2) and over a total period of 2 months.
Groups:
- Imurek®: Generic name : Azathioprine Trade name : Imurek® 50mg tablet Dosage form : Tablet containing 50 mg azathioprine Dose : 1 x Imurek 50mg Tablet per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Aspen Pharma Trading Limited, Dublin, Ireland Country of origin : Ireland
  Azathioprine: tablet
- Jayempi™: Generic name : Azathioprine
  Trade name : (Jayempi™) 10 mg/ mL Oral solution Dosage form : Oral suspension containing 10 mg/mL Azathioprine Dose : 1 x 5mL (50 mg) of Jayempi™ Oral Suspension 10mg/mL per treatment period under fasting conditions Mode of administration : Orally Manufacturer : Nova Laboratories Ltd. Country of origin : Leicester, UK
  Azathioprine: oral suspension
Arm/Group | Imurek® | Jayempi™
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imurek® (N=30) | Jayempi™ (N=30)
Headache (Nervous system disorders) | 2 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03930264/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT03930264/SAP_001.pdf